CLINICAL TRIAL: NCT02852928
Title: Orphans Unite: chILD Better Together - European Management Platform for Childhood Interstitial Lung Diseases / chILD-EU - International Register and Biobank for Children´s Interstital Lung Disease
Brief Title: European Management Platform for Childhood Interstitial Lung Diseases - chILD-EU Register and Biobank
Acronym: chILD-EU
Status: Recruiting | Type: Observational
Sponsor: Matthias Griese (Other)
Responsible Party: Sponsor-Investigator, Matthias Griese, Prof. Dr. med., Ludwig-Maximilians - University of Munich
Organization: Ludwig-Maximilians - University of Munich (Other)
Other Study IDs: chILD-EU
Record Dates: First submitted 2016-07-29; First posted 2016-08-02 (Estimated); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Lung Diseases, Interstitial; Pulmonary Alveolar Proteinosis; Pulmonary Eosinophilia; Pulmonary Fibrosis; Respiratory Distress Syndrome, Newborn; Child
Keywords: ILD; chILD
MeSH Terms: conditions — Lung Diseases, Interstitial; Pulmonary Alveolar Proteinosis; Pulmonary Eosinophilia; Pulmonary Fibrosis; Respiratory Distress Syndrome, Newborn

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Generation of a common European database and biobank Continous assessment and implementation of guidelines and treatment protocols Establishment of a large observational cohort of chILD patients Determination the value of outcomes used in child Assess treatment variations used, deliver data from defined protocols and linked outcomes

DETAILED DESCRIPTION:
Objective 1: Generation of a common European database and biobank. The existing national programmes to collect data on chILD in three countries (France, Germany, UK) will enable the consortium to swiftly adapt current frameworks to a functionally appropriate pan-European web-based database and biobank. Importantly, compatibility with ongoing United States chILD data base developments will be factored in.

Objective 2: Continuous assessment and implementation of guidelines and treatment protocols. Our Standards Working Group will convene regularly. Initial tasks will establish (a) specific diagnostic pathways, including detailed protocols for gathering clinical information, blood testing, imaging and pathology ("Best Practice Checklist"); (b) international panels of clinicians, geneticists, radiologists and pathologists who will review every diagnosis to quality control the data; and (c) detailed protocols for follow up to generate natural history data.

Objective 3: Recruitment of a carefully characterized cohort of chILD patients. European wide recruitment and interdisciplinary critical peer review of all diagnoses submitted from across Europe is imperative. Each case will be given a diagnosis independently; if no firm diagnosis is possible, we will review the case periodically as new information becomes available. During the first year of the study, clinicians´ decisions according to local practice and outcomes will be independently monitored and assessed.

Objective 4: Determine the value of outcomes used in chILD. We will systematically optimize and clarify the relative weight of a large spectrum of single and composite clinical outcomes (using both clinician and carer scoring), sequential limited chest CT (to minimise radiation exposure), lung function testing, histopathological categorization of lung biopsies, serum markers and genetic tests. Variability, reproducibility and the effects of training on reading images will be investigated.

Objective 5: Assess treatment variations used, deliver data from defined protocols and linked outcomes. This project will analyse in detail treatment and outcomes within and between subjects using data collected. Analysis of the collected data will enable us to support the definition of trial protocols planned in the future.

ELIGIBILITY:
Inclusion Criteria:

* all children with suspected or
* verified diagnosis of ILD or
* masquerading as ILD and
* those with rare localized parenchymal lung diseases

Exclusion Criteria:

* other indication as inclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 400 prevalent patients with childhood interstitial lung disease (chILD) in Europe 100 incident chILD cases per year
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2013-12 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Included subjects with specific diagnosis | 10 years
  Number of recruited subjects

SECONDARY OUTCOMES:
Survial | 10 years
  Survival of the participants

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Griese, Prof., Study Chair — Klinikum der Universität München, Dr. von Haunersches Kinderspital
Locations (3):
- Medizinische Hochschule Hannover, Hanover, Lower Saxony, Germany
- Hacettepe University, Medical Faculty, Ankara, Sihhiye, Turkey (Türkiye)
- University of Edinburgh, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Griese M, Seidl E, Hengst M, Reu S, Rock H, Anthony G, Kiper N, Emiralioglu N, Snijders D, Goldbeck L, Leidl R, Ley-Zaporozhan J, Kruger-Stollfuss I, Kammer B, Wesselak T, Eismann C, Schams A, Neuner D, MacLean M, Nicholson AG, Lauren M, Clement A, Epaud R, de Blic J, Ashworth M, Aurora P, Calder A, Wetzke M, Kappler M, Cunningham S, Schwerk N, Bush A; the other chILD-EU collaborators. International management platform for children's interstitial lung disease (chILD-EU). Thorax. 2018 Mar;73(3):231-239. doi: 10.1136/thoraxjnl-2017-210519. Epub 2017 Oct 22. PMID 29056600
- See also: chILD-EU project website — http://childeu.net